CLINICAL TRIAL: NCT04539015
Title: Randomized Study to Evaluate the Efficacy of Applying Prevena Plus to Closed Surgical Incision in Patients Undergoing CAWR and Other Laparotomy Procedures vs SOC Surgical Incision Dressing in Preventing SSI
Brief Title: Assess the Efficacy of Prevena Plus vs SOC to Closed Incision in Pts Undergoing CAWR and Other Laparotomy Procedures.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: New York Medical College (Other)
Collaborators: Acelity (Other)
Responsible Party: Principal Investigator, Rifat Latifi, Professor, General surgery, New York Medical College
Other Study IDs: 14072
Record Dates: First submitted 2020-08-13; First posted 2020-09-04 (Actual); Last update posted 2020-09-04 (Actual); Status verified 2020-08

CONDITIONS: Hernia
MeSH Terms: conditions — Hernia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group-I: Patients randomized to the Group-I will receive PREVENA Plus, which is currently being used at our institution (Prevena, KCI) and it is FDA-approved device. Dressings will be applied under sterile conditions at the end of the surgery while still in the operating room and will continuously apply for 5 days.
  Interventions: Device: Prevena Plus
- Group-II: Subjects randomized to SOC surgical incision dressing arm will receive SOC dressing for 4 days immediately following surgery. The closed incision will be covered with materials which may include sterile gauze pieces, surgical tape and tegaderm.
  Any material used for the SOC dressing will be documented.

INTERVENTIONS:
Device: Prevena Plus — PREVENA Plus is a negative pressure wound therapy device intended for use on surgical incisions that continue to drain following sutured or stapled closures.
  Groups: Group-I

SUMMARY:
The goal of this study to establish the efficacy of Prevena™ Plus in preventing surgical site infection after complex abdominal wall procedures and major laparotomies as compared to SOC dressing. We hypothesized that use of Prevena Plus will significantly decrease the incidence of Surgical Site Infection (SSI) and subsequently may have an impact over reducing hospital cost. Study data will be analyzed for clinical outcomes through 30 days. The patients will be followed every day during the hospital stay and study follow-up visits will be conducted in the clinic at 2 weeks and 1 month from the date of discharge.

DETAILED DESCRIPTION:
Background:

Postoperative wound complications are a frequent cause of surgical morbidity and a large-scale health problem. Surgical site infection leads to excess morbidity, prolonged hospitalization and increased strain on healthcare resources. It is estimated that the total annual cost for hospital-acquired infections was $9.8 billion, with SSIs contributing 33.7% to overall cost (approximately $20,785 per case). Patients undergoing major laparotomy such as elective colorectal procedures, bowel resections, solid organ tumor resection and complex abdominal wall repair (CAWR) are at high risk of developing wound complications. As a tertiary care teaching hospital, the volume of surgical cases is high which includes but not limited to Complex Abdominal wall reconstruction (CAWR) with biological mesh, elective colorectal procedures, solid organ tumor resection and organ transplant.

Investigators have started using Prevena™ incision management system over primarily closed surgical incision after all the above mentioned procedures and subjectively observed the decrease in surgical site infection.

Study Design:

This is a Prospective, Randomized, Controlled study to evaluate the efficacy of applying Prevena Plus to closed surgical incision in patients who had or undergone Complex Abdominal Wall Reconstruction with biological mesh and other major laparotomies (treatment Group) as compared to Standard of Care (SOC) surgical incision dressing (dry sterile dressing/gauze, steri-strips) in preventing surgical site infection.

Study Procedures:

Screening/Baseline: The subjects who are scheduled and or admitted at our institution for complex abdominal wall reconstruction procedure with biological mesh and other major laparotomies will be screened for eligibility to participate in the study and screening will start whenever patient comes for pre-operative visit usually 1- 3 weeks prior to and including the day of surgery. If patient agrees to participate in the study and signs the consent he/she will be randomized in the study intra-operatively. Baseline information like past medical history, past surgical history, comorbid conditions, concomitant medications, will be collected and subjects will be asked to complete the questionnaires at screening visit.

After signing the consent form, subjects will be assigned a unique, consecutive screening number for screening log tracking purposes and the screening log will also include reason for screen failure. Screening log will be filed in regulatory binder.

Screen Failure: Any eligible patient who met all the inclusion criteria and signed the consent to participate in the study but later decides not to participate in the study or if they meet any of the intra-operative exclusion criteria, randomization will not be performed and they are considered as screen failures. There will be no further study related contacts with these patients.

Randomization:

Randomization will occur intra-operatively after surgical incision closure and after confirmation of all the intra-operative inclusion criteria and none of the intra-operative exclusion criteria are met. After subjects have been assessed for eligibility and randomized in the study, they will be randomly allocated to any one of the groups in the ratio of 1:1. Randomization means that the researcher does not control which subject gets put in which group. Each participant has an equal chance of being assigned to each group. The participant will be assigned to a group by chance to eliminate bias.

Group assignments will be contained in sequentially numbered, opaque, sealed envelopes to conceal allocation from participants and investigators. Each subject will be provided with unique four digit number (1001 etc) so the data that is collected during the study participation will be saved under that unique four digit number. Once a subject number is assigned, it is not re-assigned to another subject. If subject is randomized but does not receive study treatment, he/she will be withdrawn from the study and the enrollment log will be completed with assigned subject number and includes reason for withdrawal. Enrollment log will be filed in regulatory binder.

Group I: Study Intervention: Subjects will receive PREVENA Plus after surgery and will apply for at least 5 days.

Group II: Standard of Care (SOC): Postoperative Surgical incision dressing (dry sterile dressing/gauze, steri-strips) which is currently the standard of care at our institution.

Study Intervention

Group-I subjects:

Patients randomized to the Group-I will receive PREVENA Plus, which is currently being used at our institution (Prevena, KCI) and it is FDA-approved device. Dressings will be applied under sterile conditions at the end of the surgery while still in the operating room and will continuously apply for 5 days.

Duration of Prevena Plus Therapy

• Continuously applied up to 5 days (removed earlier if there is a suspicion for wound infection or bleeding).

Group-II: Standard of Care Dressing Subjects randomized to SOC surgical incision dressing arm will receive SOC dressing for 4 days immediately following surgery. The closed incision will be covered with materials which may include sterile gauze pieces, surgical tape and tegaderm.

Any material used for the SOC dressing will be documented.

Duration of Study Participation:

* Screening: starts at Pre Admission Testing visit and includes day of surgery (subjects undergoing elective or emergent procedures).
* Treatment Duration:

  * Prevena Group: 5 days
  * SOC Group: 4 days
* Follow-up Phase: After randomization -Day 0 through 30 days (+ 7days).

Research Subject Population:

Number of Subjects Approximate number of subjects to be enrolled in this study is 170 (85 in each group).

Gender of Subjects There will be no gender based restrictions for this study.

Age of Subjects Adults 18 years of age and above will be included in this study.

Racial and Ethnic Origin There will be no enrollment restrictions based upon race or ethnic origin

Data Collection Time Periods Data will be gathered from the patients and the medical record. Data will be collected on factors such as medical history, comorbid conditions, prior surgeries, pre-operational factors, surgical technique, functional status and other items as indicated in the data collection form. This data collection will be broken down into three main time periods.

Preoperative:

Demographics: age and gender Social History: recreational drug use, smoking and alcohol. Vitals: systolic blood pressure (SBP), diastolic blood pressure (DBP), heart rate (HR), temperature (temp), respiratory rate (resp. rate), height, weight and BMI (body mass index) Lab reports: the lab tests that are done as standard of care during the hospital stay will be collected. The following lab values will be collected for the study only if they are available in subject's medical record: hemoglobin, hematocrit, white blood count (differential), sodium, BUN (blood urea nitrogen), lactate, pH, glucose, creatinine, platelet count, serum albumin, coagulation profile (PT (prothrombin time)/PTT (partial thromboplastin time) /aPTT (activated partial thromboplastin time), if available, cultures from blood, urine, sputum, trachea, wound and peritoneal fluid will be collected as well.

Comorbid Conditions: Obesity, history of Diabetes, chronic obstructive pulmonary disease (COPD), Cardiac disease, malignancy, solid organ transplant, peripheral vascular disease, cerebrovascular accident, immunosuppression, functional dependency, cirrhosis, history of acute or chronic renal failure, cirrhosis, ascites and nutritional status.

Concomitant Medications: all medications including antimicrobial medications that the subject is taking from the time subject signed the informed consent through the duration of the study.

Intraoperative:

Duration of surgery: start time and end time Amount and type of fluids Received: IV fluids and blood products received General: ASA score, Number of drains, planned/unplanned procedures and amount of blood loss Type of surgery and technique: Investigators will note the type and placement of incision , measurements of the incision, location of the mesh placement (sublay, underlay, overlay or bridge), size of mesh in cm2, anterior/posterior component separation, number of drains placed, setting of surgery (elective vs emergent/urgent).

Postoperative:

Plan for monitoring heart rate and blood pressure:

As per standard of care, if a patient is in the intensive care unit blood pressure and heart rate is monitored every hour. If patient is on the floor heart rate and blood pressure is monitored every 4hours. Arrhythmia is monitored by placing a multi-lead electrocardiogram (ECG) on the patient. As long as monitoring for arrhythmia is not hindered in any way, having a PREVENA dressing on the body does not pose any risk to the patient. Since this study does not involve any Cardiothoracic procedures and positioning of multi lead ECG for monitoring of Arrhythmias will not pose any risk to the patients. Arrhythmia is not a contraindication or a non-indicated application, it's more of PREVENA dressing placement issue when other interventions are necessary.

General: date of discharge, time of discharge, hospital length of stay, intensive care unit length of stay, (ICU LOS), ventilator days, transfer back to ICU, time of drain removal and mortality Complications: any of these postoperative complications will be collected and reported based on Clavien-Dindo classification- wound infection, Pneumonia, MI, stroke, Seroma, fistula, sepsis, urinary tract infection, venous thrombosis, pulmonary embolism, adult respiratory distress syndrome, and paralytic ileus. Post-operative seroma will be noted and documented according to Morales-Conde classification.

Investigators will also note other surgical site occurrence (SSO) dehiscence: primary and secondary. Surgical site infection: superficial and deep SSI-purulent drainage from incision, fluid accumulation, purulent fluid that is drained or positive culture with signs/symptoms.

Organism isolated from aseptically obtained culture of fluid or tissue, antimicrobials, Percutaneous or open drainage by surgeon. Debridement, hospital and ICU length of stay Disposition: home, acute rehabilitation center or subacute rehabilitation center.

Study Follow-up Visits Duration of the study is 30 days and all the follow-up visits are standard of care. Wounds will be assessed postoperatively at regular intervals until wound healing is achieved. This will occur at 2 weeks and 4 weeks after surgery, which are standard intervals in our current postoperative protocol. Investigators will analyze stitch line, pain at the incision site, any evidence of surgical site occurrence such as infection, necrosis, seroma, bulge or recurrence. All enrolled subjects are in the study for only 4 weeks and after that there will be no additional study visits but patients randomized to group-I or group-II will be followed in the clinic regularly per standard of care.

End of the Study: Study will end after the last enrolled subject completes the 30 day follow-up visit and the final study report will be submitted to IRB after manuscript or other publications are submitted and accepted.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female, 18 years of age or older
* Open abdominal wall reconstruction with biological mesh, elective colorectal procedures, solid organ tumor resection, liver transplant and elective bowel resections.
* Surgical incision closed with staplers or sutures.
* Able to provide informed consent
* Willing and able to return for scheduled study visits
* Female of child bearing age, must be negative on urine pregnancy test.
* Center for disease control (CDC) wound class I and II.
* Intra-operative inclusion criteria:
* Subject meets below criteria are eligible for randomization:
* Subject continues to meet all pre-operative inclusion criteria
* Has been classified as CDC wound Class I or II resulting in a closed surgical incision and will be able to cover the surgical incision by Prevena Plus

Exclusion Criteria:

* Age less than 18 years
* Wound left to close by secondary intention.
* Open wounds or dehisced wounds.
* Patient has known allergy or hypersensitivity to silver or adhesive tape material (acrylic compounds).
* Patients having known systemic bacterial or fungal infection at the time of surgery and local SSI before surgery. (Untreated or inadequately treated infection)
* Inadequate hemostasis of the incision
* Cellulitis of the incision area
* Subject who, in the investigator's opinion, would have any clinically significant condition that would impair his/her ability to comply with the study procedures
* Laparoscopic surgery.
* Patients undergoing perforation or diverticulitis will be excluded from the study.
* Intra-operative inclusion criteria:
* Subject who meets below intra operative criteria are considered as screen failures and are not eligible for randomization:
* If Subject meets any of the above exclusion criteria
* Subject determined to have Class III or IV wound classification procedure like open, fresh, accidental wounds, and /or major breaks in sterile technique or gross spillage from GI tract or old traumatic wounds retained devitalized tissue and those that involve existing clinical infection or perforated viscera.
* Patients who have very fragile skin around the incision are not included in the study
* If patients have any known bleeding disorders or if they refuse blood transfusions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are scheduled and or admitted at Westchester Medical Center to undergo complex abdominal wall reconstruction with Biomesh and other major laparotomies will be identified by the study staff
Sampling Method: Probability Sample
Enrollment: 170 (Estimated)
Dates: Start 2020-07-09 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2023-02-28 (Estimated)

PRIMARY OUTCOMES:
surgical site infection | 30 days
  wound infection, seroma and wound dehiscence.

SECONDARY OUTCOMES:
Hospital Admissions | 30 days
  Frequency of hospital admissions and cost

CONTACTS AND LOCATIONS:
Overall Officials: Rifat Latifi, MD, Principal Investigator — Chairman Department of Surgery
Locations (1):
- Westchester Medical Center, Valhalla, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided
No Plan.